CLINICAL TRIAL: NCT07084792
Title: Dynamic Motor Cortical Responses to Subdural Electrical Stimulation.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team is no longer moving forward with this study.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00142103
Record Dates: First submitted 2025-06-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Parkinsons Disease (PD)
Keywords: Parkinsons
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects will undergo stimulation with the device (Experimental)
  Interventions: Device: Direct cortical stimulation

INTERVENTIONS:
Device: Direct cortical stimulation — Stimulation

SUMMARY:
The purpose of this study is to better understand how subdural electrical stimulation of the brain affects motor cortical oscillations

DETAILED DESCRIPTION:
Direct cortical stimulation (DCS) has shown the potential to improve symptoms in patients with Parkinson's disease, however its effects have not been consistent in randomized studies to date, limiting widespread adoption of this technology. A critical gap in our knowledge is a detailed understanding of how DCS affects motor areas in the brain. Investigators propose using subdural DCS (sDCS) while simultaneously recording directly from motor cortex using subdural electrocorticography (sECoG) in patients undergoing deep brain stimulation surgery. Investigators expect this novel approach to broaden our understanding of sDCS application and possibly lead to therapeutic advances in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD and consented and scheduled for DBS surgery with the PI
* Age 18-80

Exclusion Criteria:

* Patients unable to actively participate in the consent process physically and/or cognitively
* Previous adverse reaction to Keppra (levetiracetam)
* Prior intracranial surgery with the exception of deep brain stimulation surgery
* Prior brain radiotherapy
* Prior history of intracranial tumor, intracranial infection or cerebrovascular malformation
* Prior history of seizures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-16 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Number of arm movements in 60 seconds | 60 seconds
  Number of arm movements in 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Rowland, M.D., Ph.D., Principal Investigator — Medical University of South Carolina